CLINICAL TRIAL: NCT00505648
Title: Treatment of DRESS (Drug Reaction With Eosinophilia and Systemic Symptoms) With Tegeline®
Brief Title: Treatment of Hypersensitivity Syndrome (DRESS) With Tegeline® (Human Immunoglobulin)
Acronym: DRESS2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Side effects valuation
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/077/HP
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Drug Hypersensitivity
Keywords: Hypersensitivity; Syndrome; Tegeline
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tegeline® — 2g/kg in IV on 2days 2g/kg in IV on 4days for patients with renal insufficiency or 65 years old.

SUMMARY:
Efficacy and tolerance of Tegeline® treatment in hypersensitivity syndrome. Immunological study of the T cell index phenotype and functionality in hypersensitivity syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Cutaneous and/or mucous eruption
* Polyadenopathy
* Body temperature > 38°C
* Hematology disorders : Hypereosinophily > 1.5 G/l, lymphocytosis > 5G/l, atypical blood lymphocytes
* Consent obtained from patient

Exclusion Criteria:

* Age < 18
* No consent obtained from patient
* IgV allergy
* Dress with very sérious visceral attack and vital diagnostic (sharp cardiac insufficiency, sharp respiratory insufficiency, hepatic insufficiency, sharp renal insufficiency)
* Oral therapy or immunosuppressive therapy (Methotrexate, cyclosporine, cyclophosphamide, etc.)
* IgA deficiency,
* MCI >=35
* Sharp renal insufficiency before Dress with creatinaemia < 60 ml/min (Cockroft)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
express healing of visceral attacks, healing of polyadenopathy and body temperature, biological abnormal values normalisation, express healing of cutaneous and mucous diseases immunological study of the T cell index phenotype | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, MD-PHD, Principal Investigator — Clinique Dermatologique - Hôpital Charles Nicolle
Locations (2):
- France (2):
  - UH-rouen, Rouen, Seine maritime
  - JOLY, Rouen